CLINICAL TRIAL: NCT02357264
Title: Thoracic Ultrasonography for the Assessment of Pulmonary Edema in Patients With Pre-Eclampsia
Brief Title: Thoracic Ultrasonography for Pulmonary Edema in Patients With Pre-Eclampsia
Status: Completed | Type: Observational
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Other Study IDs: 2014-11-25
Record Dates: First submitted 2015-01-31; First posted 2015-02-06 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2016-09

CONDITIONS: Pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pre-eclampsia: Ultrasound of Pregnant Females 18+ with pre-Eclampsia
  Interventions: Device: Ultrasound
- No pre-eclampsia.: Ultrasound of Pregnant Females 18+ with no pre-eclampsia
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound of the chest for the detection of fluid in the lung

SUMMARY:
This project will study the use of ultrasound of the chest for the detection of fluid in the lungs in patients with pre-eclampsia vs pregnant patients without pre-eclampsia. Pre-eclampsia is a syndrome usually diagnosed in the second half of pregnancy in which patients develop elevated blood pressure and may develop protein in their urine, neurologic abnormalities, fluid in the lungs, and abnormal blood tests associated with the liver and kidney. Pulmonary edema (fluid in the lungs) in pre-eclampsia can lead to patient discomfort and significant morbidity and mortality. It can be detected using chest x-ray, although this type of imaging offers significant disadvantages, including radiation, which is of particular concern in pregnant patients. In addition, previous studies have demonstrated that chest x-ray is not very accurate in the detection of fluid in the lungs. Multiple previous studies have demonstrated the utility of chest ultrasonography in detecting fluid in the chest, although the vast majority of these studies involved patients with acute decompensated heart failure. Our goal is to evaluate bedside ultrasound of the chest in patients with pre-eclampsia in comparison to normal pregnant patients to determine whether these patients have abnormal fluid in the chest.

The investigators will divide our patients into two groups. In the study group, the investigators will include patients with pre-eclampsia with or without shortness of breath, and in the control group, the investigators will include pregnant patients without pre-eclampsia. Informed consent will be obtained from all patients enrolled in the study. These patients will then undergo an ultrasound of the chest, performed by a member of the Emergency Medicine Ultrasound Division. The images will be transmitted wirelessly from the ultrasound machine to a secure web based cloud (Q-path) and will be subsequently reviewed by expert reviewers.

DETAILED DESCRIPTION:
This project will compare the use of ultrasound of the chest for the detection of fluid in the lungs in patients with pre-eclampsia vs pregnant patients without pre-eclampsia. Patients admitted to the obstetrical service will be recruited for study enrollment. We will divide our patients into two groups. In the study group, we will include patients with pre-eclampsia with or without shortness of breath, and in the control group, we will include otherwise healthy pregnant patients. We will exclude patients who are in labor or who are undergoing induction. Informed consent will be obtained from all patients enrolled in the study.

Study subjects will then undergo an ultrasound of the chest, performed by a member of the Emergency Medicine Ultrasound Division, who have experience in performing lung ultrasounds. Both hemithoraces will be divided into 4 zones: anterior inferior, anterior superior, lateral inferior, and lateral superior. Each zone will be assessed for the presence of B-lines. For a zone to be considered "positive" for pulmonary edema, there should to be a minimum of 3 B-lines. To diagnose a patient with pulmonary edema, at least two zones in both hemithoraces must be positive. The study investigator will document the presence of B-lines in each particular zone on the data collection sheet. Brief representative video clips will be recorded for each zone.

After completing the sonographic examination, the images will be transmitted wirelessly from the ultrasound machine to a secure web based cloud (Q-path) and will be subsequently interpreted by expert reviewers who will be blinded to any clinical information about the patient. They will also document their findings on a separate data collection sheet.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years of age
* Met criteria for pre-eclampsia as per ACOG guidelines for the study group
* Consent to participate in study
* Single intrauterine pregnancy

Exclusion Criteria:

1. Other cardiovascular or pulmonary problems
2. Other obstetrical or uteroplacental problems - abruption placenta, coagulopathy, immunological disorders.
3. Patients who are in labor or are received induction medications such as Pitocin.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant Females
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Dickman, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hutcheon JA, Lisonkova S, Joseph KS. Epidemiology of pre-eclampsia and the other hypertensive disorders of pregnancy. Best Pract Res Clin Obstet Gynaecol. 2011 Aug;25(4):391-403. doi: 10.1016/j.bpobgyn.2011.01.006. Epub 2011 Feb 18. PMID 21333604
- [Background] Dennis AT, Solnordal CB. Acute pulmonary oedema in pregnant women. Anaesthesia. 2012 Jun;67(6):646-59. doi: 10.1111/j.1365-2044.2012.07055.x. Epub 2012 Mar 15. PMID 22420683
- [Background] Sciscione AC, Ivester T, Largoza M, Manley J, Shlossman P, Colmorgen GH. Acute pulmonary edema in pregnancy. Obstet Gynecol. 2003 Mar;101(3):511-5. doi: 10.1016/s0029-7844(02)02733-3. PMID 12636955
- [Background] Bamfo JE, Kametas NA, Nicolaides KH, Chambers JB. Maternal left ventricular diastolic and systolic long-axis function during normal pregnancy. Eur J Echocardiogr. 2007 Oct;8(5):360-8. doi: 10.1016/j.euje.2006.12.004. Epub 2007 Feb 23. PMID 17321800
- [Background] Young P, Johanson R. Haemodynamic, invasive and echocardiographic monitoring in the hypertensive parturient. Best Pract Res Clin Obstet Gynaecol. 2001 Aug;15(4):605-22. doi: 10.1053/beog.2001.0203. PMID 11478818
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Lichtenstein D, Goldstein I, Mourgeon E, Cluzel P, Grenier P, Rouby JJ. Comparative diagnostic performances of auscultation, chest radiography, and lung ultrasonography in acute respiratory distress syndrome. Anesthesiology. 2004 Jan;100(1):9-15. doi: 10.1097/00000542-200401000-00006. PMID 14695718
- [Background] Lichtenstein D, Meziere G, Biderman P, Gepner A, Barre O. The comet-tail artifact. An ultrasound sign of alveolar-interstitial syndrome. Am J Respir Crit Care Med. 1997 Nov;156(5):1640-6. doi: 10.1164/ajrccm.156.5.96-07096. PMID 9372688

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-eclampsia | No Pre-eclampsia.
Started | 56 | 130
Completed | 56 | 130
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-eclampsia | No Pre-eclampsia. | Total
Number analyzed (Participants) | 56 | 130 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (5.93) | 31.1 (5.90) | 31.2 (5.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 130 | 186
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 56 | 130 | 186

OUTCOME MEASURES:

1. Primary Outcome: Detection of Fluid in the Lungs
Description: Detection of Fluid in the lungs in patients with pre-eclampsia vs. pregnant patients without pre-eclampsia
Time Frame: 24-36 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Pregnant Females Without Pre-Eclampsia: Pregnant Females who the OB/GYN physician suspects do not have pre-eclampsia
- Pregnant Females With Suspicion of Pre-eclampsia: Pregnant females who the OB/GYN physician has suspicion that may have pre-eclampsia
Arm/Group | Pregnant Females Without Pre-Eclampsia | Pregnant Females With Suspicion of Pre-eclampsia
Number analyzed (Participants) | 130 | 56
Participants | 2 | 3
Statistical Analysis 1: Comparison: Pregnant Females Without Pre-Eclampsia vs Pregnant Females With Suspicion of Pre-eclampsia; Test type: Other; p = .162, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Pre-eclampsia | No Pre-eclampsia.
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/130
Other Adverse Events (participants affected / at risk) | 0/56 | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes